CLINICAL TRIAL: NCT05335785
Title: Efficacy of High Intensity Lazer Therapy in Patients Diagnosed With Partial Supraspinatus Tear
Brief Title: Efficacy of High Intensity Lazer Therapy in Partial Supraspinatus Tear
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Korhan Barıs Bayram, associate professor doctor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IzmirKCU*
Record Dates: First submitted 2022-03-08; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Supraspinatus Tear
Keywords: shoulder; supraspinatus tear; rotator cuff tear; hiltherapy; lazer therapy
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 5 session lazer therapy (Active Comparator): 30 patients will be included to 5 session lazer therapy group. They will take totally 5 sessions of high-intensity laser every other day.
  Interventions: Device: High-intensity lazer therapy
- 10 session lazer therapy (Active Comparator): 30 patients will be included to 10 session lazer therapy group. They will take totally 10 sessions of high-intensity laser every other day.
  Interventions: Device: High-intensity lazer therapy
- control group (Other): 30 patients will be included to control group. They will take only exercise program three times in a week.
  Interventions: Other: Exercises

INTERVENTIONS:
Device: High-intensity lazer therapy — Patients in the laser group will be given hiltherapy (high-intensity laser) with the HIRO 3 device every other day. One session of laser therapy application consists of 3 phases: the beginning, the middle and the ending phase. The initial phases are fast scanning and the ending phase is slow scanning. A total of 2000 J will be applied to the rotatorcuff muscles, the upper part of the trapezius muscle, the deltoid muscle and the pectoralis major muscle, 1000 J in the rapid scan phase and 1000 J in the finishing phase. In the middle phase, 50 J will be applied for the trigger point (hard intramuscular points that cause referred pain) in each muscle and a maximum of 500 J in total. The total dose prescribed for patients in one session will be 2500 J. Each phase will be 15 minutes on average and the session will last for 45 minutes in total. The laser probe will be applied with 90 degrees. During the application, the practitioner and the patient will have protective glasses.
  Arms: 10 session lazer therapy; 5 session lazer therapy
Other: Exercises — Exercise program including Codman, Range of motion and streightening exercises three times in a week.
  Arms: control group

SUMMARY:
Rotatorcuff lesions constitute 10% of the causes of shoulder pain. Supraspinatus tear is one of the common rotatorcuff lesions. It affects the quality of life negatively and causes loss of range of motion and muscle strength. It can be seen due to traumatic or degenerative causes. Its incidence increases with advanced age. While the incidence was reported as 4% in the population aged 40-60 years, this rate was reported to be 17-50% in the group over the age of 60 and 80% in the group over the age of 80. Radiologically, classification is made as partial or full-thickness tears. Rotatorcuff tears can be treated conservatively or surgically. Although the risk of post-surgical rupture is reduced with new methods, the lack of desired tendon healing has led to the search for alternative applications such as biological augmentation and high-intensity laser. The aim of this study is to reveal the effectiveness of high-intensity laser therapy in patients with partial supraspinatus tear.

DETAILED DESCRIPTION:
90 patients aged 20-60 years who were diagnosed with partial supraspinatus tear and met the inclusion criteria of the study will be included in the study. Patients will be randomized into three groups: 30 patients in the first group who have 5 sessions of high-intensity laser, 30 patients in the second group who have 10 sessions of high-intensity laser, and 30 patients in the third group control group who have only exercises. It was planned to give 5 sessions of laser+exercise every other day to the the first group, 10 sessions of laser+exercise every other day to the second group, and only exercise program three days in a week to the control group. All groups will be evaluated with joint range of motion (ROM) (measurements including abduction, adduction, flexion, extension, internal and external rotation by goniometer according to neutral 0 position), visual analog scale (VAS), shoulder pain dissability index, quickdash, constant score at 0th month, 1st month, 3rd and 6th months.

ELIGIBILITY:
Inclusion Criteria:

* age between 20-65 years
* Patients with VAS>4 pain in the shoulder for at least 3 months
* Patients with at least 25% loss in the range of motion of the joint compared to the contralateral side, especially in abduction and external rotation, or on physical examination or positivity of at least one of the impingement tests including jobb, lift off, ERLS , speed, yergeson, O Brien's test, dropparm tests or popeye signs.
* Diagnose of partial supraspinatus with ultrasound or MR

Exclusion Criteria:

* Patients with incomplete skin integrity, hyperemia, signs of infection or tattoos
* Patients with suspected full-thickness tear
* History of rheumatic disease (rheumatoidarthritis, osteoarthritis, PMR)
* Patients with accompanying shoulder pathology such as calcifictendinitis
* History of malignancy
* Surgery, manipulation, mobilization, arthroscopy performed on the affected shoulder
* Steroid, local anesthetic, hyaluronic acid injection, cnesiotaping or neural therapy in the affected shoulder in the last 3 months
* Reflex sympathetic dystrophy, neurodeficit in the affected extremity
* Diabetes patients or any Patients who cannot feel the burning pain due to a peripheral neuropathy or sensory defect
* Patients with epilepsy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-12-02 (Estimated); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
VAS (visuel analog score) | 3rd month
  evaluation of pain with scale of between 0 and 10 that means 0 no pain and 10 too much pain.

SECONDARY OUTCOMES:
Constant score | 6 th month
  The Constant score (CS) is one of the most frequently applied tools for the assessment of the shoulder joint.The Constant score is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Korhan Barış Bayram, assoc. prof., Study Director — Katip Celebi University
Locations (1):
- Izmir Katip Celebi University, Izmir, Karabaglar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
study protocol will be shared for first 6 months after the study finish results and statisitcs will be shared.
Supporting Information: Study Protocol
Time Frame: when the study start and data will be avaliable for 6 months
Access Criteria: study protocol will be shared for first 6 months after the study finish results and statisitcs will be shared.

REFERENCES:
- [Background] Meislin RJ, Sperling JW, Stitik TP. Persistent shoulder pain: epidemiology, pathophysiology, and diagnosis. Am J Orthop (Belle Mead NJ). 2005 Dec;34(12 Suppl):5-9. PMID 16450690
- [Background] Boileau P, Brassart N, Watkinson DJ, Carles M, Hatzidakis AM, Krishnan SG. Arthroscopic repair of full-thickness tears of the supraspinatus: does the tendon really heal? J Bone Joint Surg Am. 2005 Jun;87(6):1229-40. doi: 10.2106/JBJS.D.02035. PMID 15930531
- [Background] Elsodany AM, Alayat MSM, Ali MME, Khaprani HM. Long-Term Effect of Pulsed Nd:YAG Laser in the Treatment of Patients with Rotator Cuff Tendinopathy: A Randomized Controlled Trial. Photomed Laser Surg. 2018 Sep;36(9):506-513. doi: 10.1089/pho.2018.4476. PMID 30188253
- [Background] Haslerud S, Magnussen LH, Joensen J, Lopes-Martins RA, Bjordal JM. The efficacy of low-level laser therapy for shoulder tendinopathy: a systematic review and meta-analysis of randomized controlled trials. Physiother Res Int. 2015 Jun;20(2):108-25. doi: 10.1002/pri.1606. Epub 2014 Dec 2. PMID 25450903
- [Background] Aleem AW, Brophy RH. Outcomes of rotator cuff surgery: what does the evidence tell us? Clin Sports Med. 2012 Oct;31(4):665-74. doi: 10.1016/j.csm.2012.07.004. PMID 23040552

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT05335785/Prot_SAP_000.pdf